CLINICAL TRIAL: NCT00517712
Title: Molecular Remission With Arsenic Trioxide in Acute Promyelocytic Leukemia: Indian APL Study Group - IAPLSG
Brief Title: Single Agent Arsenic Trioxide in the Treatment of Newly Diagnosed Acute Promyelocytic Leukemia
Acronym: IAPLSG04
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christian Medical College, Vellore, India (Other)
Collaborators: Ministry of Science and Technology, India (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAPLSG2004; BT/PR4460/Med/14/531/2003
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2007-08-17 (Estimated); Status verified 2007-08

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute promyelocytic leukemia; Arsenic trioxide; Molecular remission; Toxicity profile; Maintenance therapy
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Duration of maintenance therapy with single agent ATO of 12 months
  Interventions: Drug: Single agent arsenic trioxide
- B (Active Comparator): Duration of maintenance therapy with single agent ATO for 6 months
  Interventions: Drug: Single agent arsenic trioxide

INTERVENTIONS:
Drug: Single agent arsenic trioxide — duration of maintenance therapy, 6 months versus 12 months

SUMMARY:
There is very limited data on the use of arsenic trioxide in newly diagnosed patients with acute promyelocytic leukemia. The use of arsenic trioxide was limited to relapsed patients mainly because of the superior efficacy of ATRA as primary therapy for newly diagnosed APML. Though the early study by Niu et al showed 72% remission rates in 11 newly diagnosed patients, the role of arsenic trioxide as primary therapy was limited by the hepatic toxicity seen in this study. Studies from our centre have shown remission rates of 70-75% in newly diagnosed patients with acute promyelocytic leukemia. There was no major toxicity seen related to the administration of arsenic trioxide. Follow up data on these patients continue to show long term remission rates above 70%. These remission rates are similar to the data available in patients with acute promyelocytic leukemia treated with ATRA. Lu et al studied 19 patients treated with oral arsenic (Tetra-arsenic tetra-sulfide) wherein 84% achieved hematological remission with disease free survival of 76% at 3 years. Studies from other groups using arsenic trioxide alone or in combination with ATRA have shown similar remission rates. Arsenic trioxide as primary therapy for patients with newly diagnosed acute promyelocytic leukemia is a very attractive treatment option for developing countries mainly because of the low cost involved along with the favorable toxicity profile. However long term remission data is still not available and the ideal course and duration of treatment still needs to be defined. This multi-center study aims to further clarify the efficacy of this agent in the treatment of newly diagnosed cases of acute promyelocytic leukemia and to study the optimal maintenance regimen.

DETAILED DESCRIPTION:
This multicenter trial will study the clinical and molecular response among patients with newly diagnosed acute promyelocytic leukemia (APL) who fulfill the inclusion and exclusion criteria.

Patients included in this trial should have been diagnosed to have Acute Promyelocytic Leukemia morphologically on FAB criteria. This is sufficient to initiate therapy with arsenic trioxide (ATO) but this diagnosis has to be confirmed using either Fluorescent in situ hybridization (FISH) for t(15;17) or reverse transcriptase polymerase chain reaction assay (RT-PCR) for PML-RARalpha transcripts within 7 days of inclusion into the study.

All these patients would have in the absence of this study received only palliative therapy due to the lack of resources to support standard chemotherapy.

Women who are pregnant will not be considered for this study.

Treatment Protocol: All patients who are included in this study will be initiated on treatment with ATO. Arsenic tri-oxide (10 mg/10ml) will be diluted in 500 ml of Dextrose Saline (only glass bottles to be used) and infused intravenously over 3 - 4 hours once a day.

No premedication is required prior to administration of the drug. The dosage schedule for administration will be as follows:

Adults: 10 mg once a day Children or adults <45kg: 0.15 mg/kg/day (maximum dose = 10mg) once a day

The total courses of therapy will be as follows:

Induction therapy: Induction therapy will be continued till ANC> 1.5 x 10e9/L and Platelet count > 100 x 10e9/L along with the absence of abnormal promyelocytes in peripheral smear on 2 consecutive occasions. Once this is achieved, bone marrow studies will be done to assess remission. If the bone marrow shows < 5% of myeloblasts and promyelocytes along with a normocellular to mildly hypocellular marrow, arsenic can be stopped. If not in CR, arsenic is continued for an additional 2 weeks and a repeat bone marrow is done to confirm CR. Arsenic tri-oxide will be given for a maximum of 60 days following which the patient would be considered a non-responder/partial responder and excluded from further treatment. If bone marrow shows <5% blasts and promyelocytes at 60 days but peripheral blood count criteria for CR are not fulfilled, patient can be still be continued on the study regimen.

Consolidation therapy: All patients who achieve CR will receive consolidation therapy for a period of 28 days after an interval of 4 weeks from achieving hematological CR. The dosage and mode of administration will be similar to the schedule followed in induction.

Maintenance therapy: All patients who are in molecular CR at the end of consolidation therapy will be randomized into 2 groups:

Group A: This group will receive 12 months of maintenance therapy. ATO will be administered for 10 days every month for a period of 12 months.

Group B: This group will receive 6 months of maintenance therapy. ATO will be administered for 10 days every month for a period of 6 months.

All patients who continue to be RT-PCR positive at the end of consolidation will not be randomized and will continue to receive all the courses of maintenance treatment. Subsequent therapy will be individualized based on the molecular monitoring results.

A total of 400 patients will be recruited at the time of initiation into this study. We expect a loss to follow up/treatment failure/death of approximately 10% of the study population and hence 360 patients will be randomized into the final 2 arms of the study ie maintenance therapy for 12 months versus 6 months after completing the consolidation therapy.

Patients with CNS disease will be treated with therapeutic Radiotherapy and intrathecal chemotherapy using Cytosine, Hydrocortisone and Methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this trial should have been diagnosed to have Acute Promyelocytic Leukemia morphologically on FAB criteria. This is sufficient to initiate therapy with arsenic tri-oxide but this diagnosis has to be confirmed using either Fluorescent in situ hybridization (FISH) for t(15;17) or reverse transcriptase polymerase chain reaction assay (RT-PCR) for PML-RARalpha transcripts within 7 days of inclusion into the study.
* All these patients would have in the absence of this study received only palliative therapy due to the lack of resources to support standard chemotherapy.

Exclusion Criteria:

* Women who are pregnant
* Patients with acute promyelocytic leukemia who are found on standard karyotyping/ FISH/RTPCR to have t(11;17) or t(5;17).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-06; Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Measure complete hematological remission rate | 60 days
Measure complete molecular remission rate | 3 months
Measure duration of response | 5 years

SECONDARY OUTCOMES:
Document early and late toxicities | 5 years
Measure relapse rates | 5 years
Measure treatment related mortality | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Mammen Chandy, MD, Principal Investigator — Christian Medical College, Vellore, India
Locations (9):
- India (9):
  - Kidwai Memorial Institute of Oncology, Bangalore, Karnataka
  - St. Johns Hospital, Bangalore, Karnataka
  - Regional Cancer Center, Trivandrum, Kerala
  - Prince Aly Khan Hospital, Mumbai, Maharashtra
  - KEM Hospital, Mumbai, Maharashtra
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Institute Rotary Cancer Hospital, New Delhi, New Delhi
  - Netaji Subhash Chandra Bose Cancer Research Institute, Kolkata, West Bengal

REFERENCES:
- [Background] Mathews V, George B, Lakshmi KM, Viswabandya A, Bajel A, Balasubramanian P, Shaji RV, Srivastava VM, Srivastava A, Chandy M. Single-agent arsenic trioxide in the treatment of newly diagnosed acute promyelocytic leukemia: durable remissions with minimal toxicity. Blood. 2006 Apr 1;107(7):2627-32. doi: 10.1182/blood-2005-08-3532. Epub 2005 Dec 13. PMID 16352810
- [Background] George B, Mathews V, Poonkuzhali B, Shaji RV, Srivastava A, Chandy M. Treatment of children with newly diagnosed acute promyelocytic leukemia with arsenic trioxide: a single center experience. Leukemia. 2004 Oct;18(10):1587-90. doi: 10.1038/sj.leu.2403480. PMID 15356649
- [Background] Mathews V, Balasubramanian P, Shaji RV, George B, Chandy M, Srivastava A. Arsenic trioxide in the treatment of newly diagnosed acute promyelocytic leukemia: a single center experience. Am J Hematol. 2002 Aug;70(4):292-9. doi: 10.1002/ajh.10138. PMID 12210810
- [Background] Mathews V, Chandy M, Srivastava A. Arsenic trioxide in the management of acute promyelocytic leukaemia. Natl Med J India. 2001 Jul-Aug;14(4):215-22. PMID 11547528
- [Background] George B, Mathews L, Balasubramanian P, Shaji RV, Srivastava A, Chandy M. Molecular remission with arsenic trioxide in patients with newly diagnosed acute promyelocytic leukemia. Haematologica. 2004 Oct;89(10):1266-7. PMID 15477216
- [Background] Mathews V, Desire S, George B, Lakshmi KM, Rao JG, Viswabandya A, Bajel A, Srivastava VM, Srivastava A, Chandy M. Hepatotoxicity profile of single agent arsenic trioxide in the treatment of newly diagnosed acute promyelocytic leukemia, its impact on clinical outcome and the effect of genetic polymorphisms on the incidence of hepatotoxicity. Leukemia. 2006 May;20(5):881-3. doi: 10.1038/sj.leu.2404165. No abstract available. PMID 16525498
- [Background] Mathews V, Thomas M, Srivastava VM, George B, Srivastava A, Chandy M. Impact of FLT3 mutations and secondary cytogenetic changes on the outcome of patients with newly diagnosed acute promyelocytic leukemia treated with a single agent arsenic trioxide regimen. Haematologica. 2007 Jul;92(7):994-5. doi: 10.3324/haematol.10802. PMID 17606455